CLINICAL TRIAL: NCT01767701
Title: A Phase II Baseline Versus Treatment Study to Determine the Efficacy of Raltegravir (Isentress) in Preventing Progression of Relapsing Remitting Multiple Sclerosis as Determined by Gadolinium-enhanced MRI
Brief Title: Raltegravir (Isentress) Pilot Study in Relapsing Multiple Sclerosis
Acronym: INSPIRE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Gavin Giovannoni, Professor Gavin Giovannoni, Chair of Neurology, Queen Mary University of London
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 008717QM; 2012-004847-61 (EudraCT Number)
Record Dates: First submitted 2013-01-07; First posted 2013-01-14 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: raltegravir; MS; RRMS; Charcot Project
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Raltegravir (Experimental): All eligible patients will complete a 3 months observation period (no medications) followed by 3 months on treatment period. During the treatment period patients will be treated with open label raltegravir 400mg twice daily.
  Interventions: Drug: Raltegravir

INTERVENTIONS:
Drug: Raltegravir — 400mg twice daily for 3 months
  Other Names: Isentress

SUMMARY:
The purpose of this study is to determine whether raltegravir is effective in preventing progression of relapsing remitting multiple sclerosis as determined by gadolinium- enhanced MRI.

DETAILED DESCRIPTION:
There is accumulating research evidence that Human Endogenous Retrovirus (HERV) and herpes viruses (in particular Epstein-Barr Virus) are involved in the pathogenesis of multiple sclerosis. People with active MS have higher levels of HERVs than people either without MS or who have other neurological conditions. It has been shown that HERVs may produce neurotoxic proteins/antigens associated with MS activity and disease progression. This is the first clinical trial investigating the hypothesis that the antiretroviral drug raltegravir may suppress HERV activity and ameliorate progression of relapsing remitting MS. Raltegravir is an integrase inhibitor which blocks retroviral replication. A recent experimental study suggests that raltegravir may also be active against herpes viruses.

Eligible participants (see Inclusion/Exclusion Criteria) will be observed for 3 months having monthly brain Gadolinium enhanced MRIs and blood/urine/saliva sampling (baseline). Then they will be treated with raltegravir (one 400mg pill taken twice a day) for 3 months. During treatment period participants will continue to have monthly MRIs and blood/saliva/urine sampling. Participants will have monthly clinical and neurological examinations and they will complete questionnaires assessing response to treatment. Participants will have screening and study visits at The Royal London Hospital, Whitechapel. Monthly MRIs will be performed at the Institute of Neurology at Queens Square, London.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18-55 years of age.
* Diagnosis of MS, according to the revised McDonald Criteria 2010.
* EDSS score of 0-6.0 inclusive.
* Documented at least one relapse within the past 12 months or at least one Gd-enhanced lesion on the brain MRI detected within 3 months prior to screening date
* Gd-enhanced lesion on screening MRI (if MRI not used to meet screening criteria above).
* Female patients of childbearing potential will be expected to be on appropriate contraception (hormonal or barrier method of birth control; abstinence) from time of consent until 6 weeks after treatment discontinuation. (the repeated administration of gadolinium and MRI are not recommended during pregnancy). NOTE: Subjects are considered not of child bearing potential if they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal.
* Females of childbearing potential must have a negative urine pregnancy test prior to every MRI scan/ within 7 days prior to being registered for protocol therapy.
* Must give written informed consent and authorize the release and use of protected health information, as required by local law.
* Able and willing to undergo blood, saliva and urine sampling at regular intervals as defined by the protocol.
* Able and willing to receive Gadolinium enhanced MRI's at regular intervals as defined by the protocol.
* Able to comply with study requirements.

Exclusion Criteria:

* Pregnant or breastfeeding or unwilling to use contraception.
* Treatment with immunosuppressive, immunomodulatory or experimental treatments within the last 6 months of enrolment in the study, but excluding pulsed intravenous or oral steroids for treatment of MS relapse.
* No pulsed intravenous or oral steroids in the 30 days preceding the baseline assessment.
* Patients presenting with medical disorder deemed severe or unstable by the CI such as poorly controlled diabetes or arterial hypertension, severe cardiac insufficiency, unstable ischemic heart disease, abnormal liver function tests (>2.5 times ULN) and abnormal complete blood count (in particular leukopenia, as defined by a lymphocyte count <500, neutrophil <1.5 or platelet count < 100, or thrombocytopenia < 1.5 LLN), or any medical condition which, in the opinion of the chief investigator, would pose additional risk to the patient.
* Presence of human immunodeficiency virus antibodies.
* Patients receiving proton pump inhibitors (e.g. omeprazole/esomeprazole)
* Patients with active hepatitis B or/and C with liver function tests >2.5 times ULN
* Exposure to any other investigational drug within 30 days of enrolment in the study.
* Prior history of malignancy unless an exception is granted by the Chief Investigator.
* History of uncontrolled drug or alcohol abuse within 6 months prior to enrolment into the study.
* Patients treated with Rifampicin in past four weeks.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2013-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julian Gold, Prof, Principal Investigator — Queen Mary University of London; Gavin Giovannoni, Principal Investigator — Queen Mary University of London
Locations (1):
- The Royal London Hospital, London, United Kingdom

REFERENCES:
- [Background] Christensen T. HERVs in neuropathogenesis. J Neuroimmune Pharmacol. 2010 Sep;5(3):326-35. doi: 10.1007/s11481-010-9214-y. Epub 2010 Apr 27. PMID 20422298
- [Background] Perron H, Germi R, Bernard C, Garcia-Montojo M, Deluen C, Farinelli L, Faucard R, Veas F, Stefas I, Fabriek BO, Van-Horssen J, Van-der-Valk P, Gerdil C, Mancuso R, Saresella M, Clerici M, Marcel S, Creange A, Cavaretta R, Caputo D, Arru G, Morand P, Lang AB, Sotgiu S, Ruprecht K, Rieckmann P, Villoslada P, Chofflon M, Boucraut J, Pelletier J, Hartung HP. Human endogenous retrovirus type W envelope expression in blood and brain cells provides new insights into multiple sclerosis disease. Mult Scler. 2012 Dec;18(12):1721-36. doi: 10.1177/1352458512441381. Epub 2012 Mar 28. PMID 22457345
- [Background] Farrell RA, Antony D, Wall GR, Clark DA, Fisniku L, Swanton J, Khaleeli Z, Schmierer K, Miller DH, Giovannoni G. Humoral immune response to EBV in multiple sclerosis is associated with disease activity on MRI. Neurology. 2009 Jul 7;73(1):32-8. doi: 10.1212/WNL.0b013e3181aa29fe. Epub 2009 May 20. PMID 19458321
- [Background] Nadal M, Mas PJ, Blanco AG, Arnan C, Sola M, Hart DJ, Coll M. Structure and inhibition of herpesvirus DNA packaging terminase nuclease domain. Proc Natl Acad Sci U S A. 2010 Sep 14;107(37):16078-83. doi: 10.1073/pnas.1007144107. Epub 2010 Aug 30. PMID 20805464

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients 18-55 years of age with RRMS, as per McDonald Criteria 2010, EDSS up to 6.0, relapse within the past 12 months or at least one active Gd enhanced lesion on brain MRI within the 3 months prior to consent. All participants were recruited at the Clinical Research Centre of the Royal London Hospital and drawn from greater London.
Pre-assignment Details: 31 subjects screened. 8 had no evidence of Gd enhancing lesions in their baseline MRI and were screen failed. Of the 23 participants who were recruited into the study 3 were withdrawn prior to starting the treatment phase; one at the request of the participant and the remaining two due to MS relapse.
Period: Overall Study
Arm/Group | Raltegravir
Started | 20 (All 20 patients who entered the treatment phase completed the six months trial period.)
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Raltegravir
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 6
Region of Enrollment [Number; unit: participants]
  United Kingdom | 20

OUTCOME MEASURES:

1. Primary Outcome: The Number of New or Recurrent Gd-enhancing Lesions That Appear on Brain T1-weighted MRI
Description: Demonstrate in subjects with relapsing remitting multiple sclerosis a reduction in the number of new or recurrent Gd-enhancing lesions that appear on brain T1-weighted MRI over the period of treatment with raltegravir, compared to baseline.
  Within patient change in number of lesions was calculated by subtracting the after treatment period (3 months) minus before treatment period (3 months).
Time Frame: Baseline and at 6 months
Population: ITT
Measure: Mean (Full Range); unit: lesions
Arm/Group | Raltegravir
Number analyzed (Participants) | 20
lesions | 0.12 [-2.67 to 3.33]

2. Secondary Outcome: The Cumulative Number of New or Enlarging T2 Weighted Lesions on Brain MRI.
Description: Demonstrate a reduction in the cumulative number of new or enlarging T2 weighted lesions on brain MRI over the period of treatment with Raltegravir compared with baseline.
  Within-patient changes in lesion count calculated after-before.
Time Frame: Baseline and monthly for 6 months
Population: ITT
Measure: Mean (Full Range); unit: T2-weighted lesions
Arm/Group | Raltegravir
Number analyzed (Participants) | 20
T2-weighted lesions | 0.19 [-4.0 to 5.00]

3. Secondary Outcome: Change in Score on Multiple Sclerosis Functional Composite (MSFC). This a Composite Score Based on the Measurement of Time in Seconds for the Three Separate Measurements.
Description: Explore preliminary clinical responses in relapsing-remitting multiple sclerosis subjects treated with Raltegravir, compared with baseline as measured by Patient Reported Outcomes (Questionnaires). The MSFC is a composite score consisting of the standardly derived composite score from 9-hole peg test (9HPT), timed walk and PASAT scores. 9HPT is measured as timed speed to complete the task; higher scores indicate less disability. The 25-foot walk is measured as timed speed; higher scores indicate less disability. The Paced Auditory Serial Addition Test (PASAT) The PASAT is a measure of cognitive function that assesses auditory information processing speed and flexibility, as well as calculation ability. It is a timed speed test measured in seconds. In the PASAT a lower score indicates less disability.
Time Frame: Baseline and monthly until month 6.
Population: ITT
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Raltegravir
Number analyzed (Participants) | 20
seconds
  25 foot walking test in seconds | -0.24 (28.2)
  9 hole peg test as a timed measurement | 0.05 (0.01)
  PASAT. This is a TIMED measurement | 49.72 (8.81)

4. Secondary Outcome: Changes in Kurtzke Extended Disability Status Scale (EDSS) Score
Description: The Kurtzke Expanded Disability Status Scale (EDSS) is a method of quantifying disability in multiple sclerosis. The scale has been developed by John F. Kurtzke. The EDSS quantifies disability in eight Functional Systems (FS) and allows neurologists to assign a Functional System Score (FSS) in each of these. 0 = Normal 1-1.5 = No disability, but some abnormal neurological signs 2-2.5 = Minimal disability 3-4.5 = Moderate disability, affecting daily activities, but you can still walk. A lower score indicates less disability.
  5-8 = More severe disability, impairing your daily activities and requiring assistance with walking 8.5-9.5 = Very severe disability, restricting you to bed 10 = Death EDSS scores were measured monthly over 6 months and the mean of the measurements for the first three months (baseline) was recorded to use calculate the change from baseline compared with the mean of measurements taken monthly during the second three months (treatment).
Time Frame: Baseline and monthly to month 6
Population: All patients enrolled in clinical trial
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Raltegravir: All eligible patients will complete a 3 months observation period (no medications) followed by 3 months on treatment period. During the treatment period patients will be treated with open label raltegravir 400mg twice daily. The EDSS score is determined by the mean score over three months after treatment minus the mean score of the three months before treatment
  Raltegravir: 400mg twice daily for 3 months
Arm/Group | Raltegravir
Number analyzed (Participants) | 20
units on a scale | 2.55 (0.92)

5. Secondary Outcome: Cumulative Number of Gd-T1 Enhancing Lesions
Description: This measure is the number of gadolinium-enhancing T1 lesions as determined by MRI taken on the monthly basis during the six months of the study.
Time Frame: At Baseline and monthly for 6 months
Population: ITT
Measure: Mean (Full Range); unit: Gadolinium enhancing T1 lesions
Arm/Group | Raltegravir
Number analyzed (Participants) | 20
Gadolinium enhancing T1 lesions | 3.08 [0 to 16]

6. Secondary Outcome: Percent of Subjects With Scans Free From Enhancing Lesions in Raltegravir Treated Subjects vs. Baseline
Description: This measure is the cumulative percentage of subjects who had scans free from Gd enhancing lesions during the first three months (baseline) compared with the second three months (treatment). These percentages are expressed as a total percentage for the baseline and for the treatment periods.
Time Frame: Baseline to 6 months
Population: ITT
Measure: Number; unit: percentage of subjects
Arm/Group | Raltegravir
Number analyzed (Participants) | 20
percentage of subjects | 15

7. Other Pre Specified Outcome: Mean Number of Adverse Events Per Patient
Description: This outcome will be assessed by blood and urine sampling; collection of patient reported symptoms and neurological and physical exams.
  This measure is the total number of adverse events recorded for each type of event during the study period. The number of participants is 31 which is the number screened and enrolled in the study. Eleven participants did not meet the criterion for baseline i.e. having a gadolinium enhancing lesion on MRI at the baseline visit and therefore did not continue to the baseline observation period. The adverse events for the 11 participants who did not begin the study observation period were recorded during the screening period and added to the 20 participants who were studied during the 6 months of the study. Adverse events are recorded as total number during the study period. Each patient may have had more than one adverse event.
Time Frame: Screening to six months
Population: ITT
Measure: Mean (Full Range); unit: Adverse events
Arm/Group | Raltegravir
Number analyzed (Participants) | 31
Adverse events | 7.9 [1.0 to 22.0]

8. Other Pre Specified Outcome: Effect of Raltegravir Therapy on Specific Inflammatory Marker of MS Activity.
Description: Measured by Human C-Reactive Protein (HCRP) which is a measure of general inflammation. The higher the value the more inflammatory response is present. The HCRP was measured monthly for six months. The mean value for the baseline three months was compared with the mean value taken for the second (treatment) three months.
Time Frame: Baseline to 6 months
Population: ITT
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | Raltegravir
Number analyzed (Participants) | 20
ng/mL | 535.82 [191.25 to 7397.33]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the time patients signed the informed consent to the end of the study period, which was up to 7 months for each patient, including screening period.
Description: Adverse events were recorded from the time subjects signed the informed consent form. 31 patients signed the informed consent and 20 were eligible for enrollment in the observational and treatment phases of the study. 11 patients were deemed not eligible as they did not have active Gd-enhanced lesions during screening.
Arm/Group | Raltegravir
Serious Adverse Events (participants affected / at risk) | 1/31
Other Adverse Events (participants affected / at risk) | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raltegravir (N=31)
MS relapse (Nervous system disorders) | 1 (1) — MS relapse requiring hospitalisation for administration of IV methylprednisolone. Normal practise would not be hospital admission but the patient had no care at home and due to MS relapse could care for self at home.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raltegravir (N=31)
Adenopathies (Immune system disorders) | 2 (2)
Itchy eyes (Immune system disorders) | 1 (1)
Allergic skin rash worsening (Immune system disorders) | 1 (1)
Hayfever congestion (Immune system disorders) | 1 (1)
Hayfever worsening (Immune system disorders) | 1 (1)
Headache (General disorders) | 10 (12)
Liver function test abnormal (General disorders) | 1 (1)
Liver function test increased (General disorders) | 2 (2)
Dizziness (General disorders) | 3 (3)
Fall (General disorders) | 5 (5)
Insomnia (General disorders) | 2 (2)
Poor sleep (General disorders) | 1 (1)
Nausea (General disorders) | 2 (2)
Swelling in left arm (General disorders) | 1 (1)
Stomach pain (General disorders) | 2 (2)
Loss of libido (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Dysphonia (General disorders) | 1 (1)
Problems concentrating (General disorders) | 1 (1)
Stiff neck (General disorders) | 1 (1)
Fainting (General disorders) | 1 (1)
Vivid dreams (General disorders) | 1 (1)
Tiredness (General disorders) | 1 (1)
Night sweats (General disorders) | 1 (1)
Dry mouth (General disorders) | 1 (1)
Weight loss diet (General disorders) | 2 (2)
Lack of motivation (General disorders) | 1 (1)
Asymptomatic low blood pressure (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Choking on liquids (General disorders) | 1 (1)
Flushing to face (General disorders) | 1 (1)
Strange sensation when swallowing (General disorders) | 1 (1)
Swelling feelings in fingers (General disorders) | 1 (1)
Depression (Psychiatric disorders) | 4 (4)
Depression worsening (Psychiatric disorders) | 1 (1)
Low mood (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Panick attacks increased (Psychiatric disorders) | 1 (1)
Emotional instability (Psychiatric disorders) | 1 (1)
Menopause onset (Reproductive system and breast disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Pelvic mass (Reproductive system and breast disorders) | 1 (1)
Haematoma (Injury, poisoning and procedural complications) | 2 (2)
Bruised knee (due to fall) (Injury, poisoning and procedural complications) | 1 (1)
Broken toenail (Injury, poisoning and procedural complications) | 1 (1)
Cut knee (Injury, poisoning and procedural complications) | 1 (1)
Twisted knee (Injury, poisoning and procedural complications) | 1 (1)
Hurt wrist (Injury, poisoning and procedural complications) | 1 (1)
Hypertension (Cardiac disorders) | 4 (7)
Tachycardia (Cardiac disorders) | 1 (2)
Hypertension worsening (Cardiac disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Wheeze (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyslipidemia (Blood and lymphatic system disorders) | 10 (17)
Mycrocytic anemia (Blood and lymphatic system disorders) | 1 (1)
Hypoglycemia (Blood and lymphatic system disorders) | 1 (1)
Normocytic anaemia (Blood and lymphatic system disorders) | 1 (1)
Multiple sclerosis relapse (Nervous system disorders) | 9 (9)
Multiple sclerosis sensory relapse (Nervous system disorders) | 5 (6)
Sensory disturbance (Nervous system disorders) | 2 (2)
Fatigue (Nervous system disorders) | 4 (4)
Fatigue increased (Nervous system disorders) | 4 (4)
Migraine (Nervous system disorders) | 4 (4)
Dysaesthesia worsening (Nervous system disorders) | 1 (1)
Nystagmus (Nervous system disorders) | 1 (1)
Neuropathic pain (Nervous system disorders) | 2 (2)
Tremor in hands (Nervous system disorders) | 1 (1)
Numbness (loss of sensation) (Nervous system disorders) | 3 (3)
tremor in arms worsened (Nervous system disorders) | 1 (1)
Subjective worsening in leg weakness (Nervous system disorders) | 1 (1)
Neurologial signs worsening (Nervous system disorders) | 1 (1)
Back pain (burning sensation) (Nervous system disorders) | 1 (1)
Visaul fatigue (Eye disorders) | 1 (1)
Decreased vision (Eye disorders) | 1 (1)
Stye (Eye disorders) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 2 (2)
Defective gastro-ileal valve (Gastrointestinal disorders) | 1 (1)
Bloated abdomen (during antibiotics) (Gastrointestinal disorders) | 1 (1)
Bladder dysfunction (Renal and urinary disorders) | 3 (4)
Dysuria (Renal and urinary disorders) | 1 (1)
Bladder problems worsening (Renal and urinary disorders) | 3 (3)
Itching (Skin and subcutaneous tissue disorders) | 2 (3)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Fungal infection (Skin and subcutaneous tissue disorders) | 3 (3)
Fungal infection worsening (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Petechial purpura (Skin and subcutaneous tissue disorders) | 1 (1)
Naevus (Skin and subcutaneous tissue disorders) | 1 (1)
Scar from mole removal (Skin and subcutaneous tissue disorders) | 1 (1)
Rash on face (Skin and subcutaneous tissue disorders) | 1 (1)
Mole on toe (Skin and subcutaneous tissue disorders) | 1 (1)
Allergic rash worsening (Skin and subcutaneous tissue disorders) | 1 (1)
Pain (Musculoskeletal and connective tissue disorders) | 14 (17)
Pain worsening (Musculoskeletal and connective tissue disorders) | 2 (2)
Carpal tunnel syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Cramps in legs (Musculoskeletal and connective tissue disorders) | 1 (1)
Common cold (Infections and infestations) | 14 (21)
Urinary tract infection (Infections and infestations) | 6 (8)
Sore throat (Infections and infestations) | 5 (5)
Cough (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 3 (3)
Tooth infection (Infections and infestations) | 1 (1)
Chest infection (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes